CLINICAL TRIAL: NCT03654638
Title: The Effect of a Soy Bread Diet Intervention on Immune Function in Men With Prostate Cancer
Brief Title: Soy Bread Diet in Improving Immune Function in Participants With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OSU-12042; NCI-2018-00808 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA169363 (NIH)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I Soy Bread Intervention (Experimental): Men who are scheduled to begin androgen deprivation therapy for prostate cancer will begin an intervention to consume 2 slices of soy bread daily for approximately 20 weeks. Blood, urine and toxicity data will be collected at regularly scheduled medical oncology visits.
  Interventions: Combination Product: Dietary Intervention; Other: Questionnaire Administration
- Arm II Wheat Bread Intervention (Active Comparator): Men who are scheduled to begin androgen deprivation therapy for prostate cancer will begin an intervention to consume 2 slices of wheat bread for approximately 20 weeks. Blood, urine and toxicity data will be collected at regularly scheduled medical oncology visits.
  Interventions: Combination Product: Dietary Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Combination Product: Dietary Intervention — The dietary intervention requires men to consume 2 slices soy bread each day for 20 weeks while initiating hormone therapy
  Other Names: Dietary Modification; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I Soy Bread Intervention
Combination Product: Dietary Intervention — The dietary intervention requires men to consume 2 slices wheat bread each day for 20 weeks while initiating hormone therapy
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm II Wheat Bread Intervention
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effects of a soy bread versus a wheat bread in improving immune function in participants who are beginning a course of androgen deprivation therapy for prostate cancer. Components found in soy foods may influence the immune system in a way that may be beneficial for prostate cancer prevention and survivorship.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To precisely define the impact of soy on myeloid derived suppressor cells (MDSC) in a human model clinical trial.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (SOY BREAD): Participants consume 2 slices of soy bread daily for approximately 20 weeks in the absence of unacceptable toxicity. Concurrent with the intervention, participants will be staring androgen deprivation therapy at the direction of their medical oncologist.

ARM II (WHEAT BREAD): Participants consume 2 slices of wheat bread daily for approximately 20 weeks in the absence of unacceptable toxicity. Concurrent with the intervention, participants will be staring androgen deprivation therapy at the direction of their medical oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Have biopsy proven adenocarcinoma of the prostate (no small cell, sarcomatoid, or other rare subtypes)
* Be planning a course of at least 5 months of androgen deprivation therapy. Patients who have had androgen deprivation therapy in the past as part of salvage therapy or primary therapy, but are initiating a new course will be eligible.
* Have a testosterone concentration within normal limits.
* No neoadjuvant hormonal or chemotherapy (other clinical trials) for their prostate cancer
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Have blood, urea, nitrogen (BUN)/creatinine (Cr), liver enzymes, complete blood count (CBC), and prothrombin time (PT)/partial thromboplastin time (PTT)/international normalized ratio (INR) within normal limits
* Voluntarily agree to participate and a sign an informed consent document
* Agree to have prostate biopsy blocks provided to the study for evaluation
* Willing to discontinue all current vitamin/mineral supplements
* Not currently be taking complementary or alternative products (i.e. PC-SPES, Saw Palmetto) that target the prostate or may impact the hormonal environment
* Agree to consume a standardized vitamin and mineral supplement (provided by the study) and avoid other nutrition, dietary, or alternative medications/supplements for the duration of the study

Exclusion Criteria:

* Have an active malignancy other than prostate cancer that requires therapy
* No diagnosed hematologic malignancy
* Not currently taking steroid medications (i.e., chronic lymphocytic leukemia [CLL])
* No chronic infection (i.e., human immunodeficiency virus-positive [HIV+])
* No history of organ transplant requiring immunosuppressive medications
* History of nephrolithiasis (renal stones)
* Renal insufficiency with creatinine > 1.8, including anyone on dialysis regardless of nadir creatinine
* Have certain medical conditions. Have no history of malabsorptive disorders or other metabolic disorders requiring special diet recommendations (for example, Crohn?s disease or gluten enteropathy)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Change in peripheral blood myeloid derived suppressor cells (MDSC) | Week 0 to week 20
  A two-sample t-test will be used to compare the differences (log-transformed if necessary to improve normality).
Treatment effect on peripheral blood MDSC | Up to week 20
  Mixed-effects regression models will be used to estimate the treatment effect on peripheral blood MDSC after adjusting for covariates such as age, compliance, and weight. A condition by time (pre versus [vs.] post) interaction will be included to test for a treatment effect. A random effect will be included for each subject to account for the dependency between the pre-post measurements. Correlations (Pearson and Spearman) between measures will be evaluated to determine if positive or negative relationships exist between the measures themselves or the week 0 to week 5 differences (e.g. MSDC vs. T-cell proliferation, MDSC vs. cytokines). Model adequacy and assumptions will be evaluated via residual plots. In the event that model assumptions are violated, outcomes will be transformed or non-parametric methods will be used. Tissue MDSC will be compared using linear regression.
Treatment effects in plasma cytokines | Up to week 20
  Mixed-effects regression models will be used to estimate the treatment effect. Correlations (Pearson and Spearman) between measures will be evaluated to determine if positive or negative relationships exist between the measures themselves or the week 0 to week 5 differences (e.g. MSDC vs. T-cell proliferation, MDSC vs. cytokines). Model adequacy and assumptions will be evaluated via residual plots. In the event that model assumptions are violated, outcomes will be transformed or non-parametric methods will be used.
Treatment effects in T-cell proliferation | Up to week 20
  Mixed-effects regression models will be used to estimate the treatment effect. Correlations (Pearson and Spearman) between measures will be evaluated to determine if positive or negative relationships exist between the measures themselves or the week 0 to week 20 differences (e.g. MSDC vs. T-cell proliferation, MDSC vs. cytokines). Model adequacy and assumptions will be evaluated via residual plots. In the event that model assumptions are violated, outcomes will be transformed or non-parametric methods will be used.
Treatment effects in prostate specific antigen (PSA) | Up to week 20
  Mixed-effects regression models will be used to estimate the treatment effect.

SECONDARY OUTCOMES:
PSA response | Up to week 20
  Mixed-effects models will be used to explore treatment effects in PSA outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu